CLINICAL TRIAL: NCT01990105
Title: Treatment of Atrial Fibrillation in Finland - the FinFib 2 Study
Brief Title: Treatment of Atrial Fibrillation in Finland
Acronym: FinFib2
Status: Completed | Type: Observational
Sponsor: Finnish Cardiac Society (Other)
Collaborators: Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FCS-2013-1; R13044 (Other: The Pirkanmaa Hospital District Ethical Committee)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; anticoagulation; antiarrhythmic medication; CHA2DS2VASc score; HAS-BLED score; CHADS2 score
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with AF in the ER: All patients with ECG-diagnosed AF who attend emergency clinics for examination or treatment of arrhythmia or other cardiac diseases during the study period will be included.

SUMMARY:
FINFIB 2 is an observational investigator-driven study that seeks to examine current treatment practice for atrial fibrillation in Finland. The investigators hypothesis is that the treatment of atrial fibrillation has improved since the introduction of new antiarrhythmic drugs and anticoagulants.

DETAILED DESCRIPTION:
FINFIB 2 is an observational investigator-driven study that seeks to examine current treatment practice for atrial fibrillation (AF) in Finland. It will produce important information such as whether the introduction of the new agents has taken place in accordance with the treatment guidelines in different parts of Finland.

Working hypothesis is that the treatment of AF has improved since the introduction of new antiarrhythmic drugs and anticoagulants. However, the investigators also expect to find out that there are geographical differences in the use of these agents. The expect outcome is that the investigators will identify these differences and be able to better homogenize the treatment of AF in different parts of the country and different levels of the health care system.

The study data will be obtained in the form of a cross-section sampling over two weeks. All patients with ECG-diagnosed AF who attend emergency clinics for examination or treatment of arrhythmia or other cardiac diseases during the study period will be included. The investigators estimate the number of patients will be about 1000. Aside from background information, risk data (e.g. CHA2DS2VASc), symptoms (EHRA classification), medication, examinations and the choice of treatment, the only data recorded about each patient with AF will be date of birth and gender. The patients will be divided into four groups according to type of AF: 1. New onset AF, 2. Paroxysmal AF, 3. Persistent AF, 4. Permanent AF. The data will be obtained by the local study doctor using online, protected data collection program. The data will be stored on a secured server, which can be accessed for data entry by the investigators at the study centers. The database is not a personal data register, as identity codes will not be stored at any point and individual patients cannot be identified later through the database. Only the investigator group will have the rights to use the database.

ELIGIBILITY:
Inclusion Criteria:

All adult patients with ECG-diagnosed AF who attend emergency clinics for examination or treatment of arrhythmia or other cardiac diseases during the study period will be included.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study data will be obtained in the form of a cross-section sampling over two weeks. All patients with ECG-diagnosed AF who attend emergency clinics for examination or treatment of arrhythmia or other cardiac diseases during the study period will be included. The estimated number of patients is about 1000.
Sampling Method: Non-Probability Sample
Enrollment: 1013 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Adherence to current atrial fibrillation treatment guidelines | Data collected during the ER visit
  All patients with ECG-diagnosed AF who attend emergency clinics for examination or treatment of arrhythmia or other cardiac diseases during the study period will be included for assessment of the adherence of their treatment to current guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Raatikainen, MD, PhD, Study Chair — Heart Center Tampere Univerisity Hospital; Juha Hartikainen, MD, Principal Investigator — Kuopio University Hospital; Timo Lauri, MD, Principal Investigator — Oulu University Hospital; Mika Lehto, MD, Principal Investigator — Helsinki University Central Hospital; Markku Mäkijärvi, MD, Principal Investigator — Helsinki University Central Hospital; Juha Lund, MD, Principal Investigator — Turku University Hospital; Heikki Mäkynen, MD, Principal Investigator — Heart Center Tampere University Hospital
Locations (5):
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Penttila T, Makynen H, Hartikainen J, Hyppola H, Lauri T, Lehto M, Lund J, Raatikainen MJP; FinFib2 investigators. Antiarrhythmic drug therapy among patients presenting to emergency department with symptomatic atrial fibrillation - a prospective nationwide cohort. Scand J Trauma Resusc Emerg Med. 2017 Aug 15;25(1):81. doi: 10.1186/s13049-017-0424-7. PMID 28810904